CLINICAL TRIAL: NCT01017471
Title: Comparison Results of Carpal Tunnel Release Between Standard Incision and Limited Incision Using PSU Retractor: A Randomized Controlled Trial
Brief Title: Carpal Tunnel Syndrome Release Using PSU Retractor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52-169-11-4-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; surgery; PSU retractor; carpal tunnel syndrome who failed to conservative treatment
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- control (Experimental): carpal tunnel release using standard incision
  Interventions: Procedure: Limited incision using PSU retractor

INTERVENTIONS:
Procedure: Limited incision using PSU retractor — carpal tunnel release using limited incision with PSU retractor will be done by orthopaedic hand surgeons

SUMMARY:
The investigators study aims to evaluate both efficacy and safety of carpal tunnel release using limited incision with the PSU retractor compared to standard incision.

The investigators will do a randomized controlled trial in 60 patients with carpal tunnel release and evaluate for outcome regarding pain, VAS score, return to work time, CTS score and complications at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as carpal tunnel syndrome who failed to conservative treatment 3 months

Exclusion Criteria:

* Underlying disease such as : DM, neuropathy
* Previous wrist or hand surgery in the same side
* Previous wrist and hand trauma
* Pregnancy

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
CTS score | 1 year

SECONDARY OUTCOMES:
VAS score | 1 year
return to work time | 1 year
satisfaction score | 1 year
complication rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sunthorn Wongsiri, MD, Principal Investigator — Prince of Songkla University, Hatyai, Songkhla, Thailand
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand